CLINICAL TRIAL: NCT02666586
Title: Effects of Faba Bean Fractions as Ingredients in Novel Food Products on Glycemia, Appetite and Metabolic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: B2015:110
Record Dates: First submitted 2015-11-19; First posted 2016-01-28 (Estimated); Last update posted 2023-01-23 (Actual); Status verified 2021-04

CONDITIONS: Faba Bean; Post-prandial Blood Glucose; Appetite; Satiety Hormones; Insulin
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (5):
- Control smoothie (Placebo Comparator): Control smoothie with 32 g corn maltodextrin without added faba bean fractions.
  Interventions: Other: Faba bean powder smoothie; Other: Faba bean protein concentrate smoothie; Other: Faba bean starch smoothie; Other: Faba bean protein isolate smoothie
- Faba Bean powder smoothie (Experimental): Breakfast smoothie with 32 g whole faba bean powder.
  Interventions: Other: Faba bean protein concentrate smoothie; Other: Faba bean starch smoothie; Other: Faba bean protein isolate smoothie; Other: Non-pulse smoothie smoothie
- Faba bean protein concentrate smoothie (Experimental): Breakfast smoothie with 32 g faba bean protein concentrate.
  Interventions: Other: Faba bean powder smoothie; Other: Faba bean starch smoothie; Other: Faba bean protein isolate smoothie; Other: Non-pulse smoothie smoothie
- Faba bean starch smoothie (Experimental): Breakfast smoothie with 33 g faba bean starch.
  Interventions: Other: Faba bean powder smoothie; Other: Faba bean protein concentrate smoothie; Other: Faba bean protein isolate smoothie; Other: Non-pulse smoothie smoothie
- Faba bean protein isolate smoothie (Experimental): Breakfast smoothie with 32 g faba bean protein isolate.
  Interventions: Other: Faba bean powder smoothie; Other: Faba bean protein concentrate smoothie; Other: Faba bean starch smoothie; Other: Non-pulse smoothie smoothie

INTERVENTIONS:
Other: Faba bean powder smoothie — Breakfast smoothie with 32 g whole faba bean powder (300g).
  Arms: Control smoothie; Faba bean protein concentrate smoothie; Faba bean protein isolate smoothie; Faba bean starch smoothie
Other: Faba bean protein concentrate smoothie — Breakfast smoothie with 32 g faba bean protein concentrate.
  Arms: Control smoothie; Faba Bean powder smoothie; Faba bean protein isolate smoothie; Faba bean starch smoothie
Other: Faba bean starch smoothie — Breakfast smoothie with 33 g faba bean starch.
  Arms: Control smoothie; Faba Bean powder smoothie; Faba bean protein concentrate smoothie; Faba bean protein isolate smoothie
Other: Faba bean protein isolate smoothie — Breakfast smoothie with 32 g faba bean protein isolate.
  Arms: Control smoothie; Faba Bean powder smoothie; Faba bean protein concentrate smoothie; Faba bean starch smoothie
Other: Non-pulse smoothie smoothie — Control smoothie with 32 g corn maltodextrin without added faba bean fractions.
  Arms: Faba Bean powder smoothie; Faba bean protein concentrate smoothie; Faba bean protein isolate smoothie; Faba bean starch smoothie

SUMMARY:
To describe the effect and mechanisms of action faba bean powder and fractions (protein, starch and fiber) on glucose and insulin homeostasis, food intake, satiety and metabolic regulation in young adults (18 to 30 years).

DETAILED DESCRIPTION:
The overall objective is to describe the effect and mechanisms of action of faba bean powder and fractions (protein, starch and fiber) on glucose and insulin homeostasis, food intake, satiety and metabolic regulation in young adults (18 to 30 years). The specific objectives are to test the acute effects of different faba bean ingredient smoothie on: 1) post-prandial blood glucose, appetite, satiety hormone and insulin for 200 minutes, and 2) food intake 120 minutes following consumption of the faba bean smoothie. Two short-term acute studies will be conducted to meet these objectives. Both acute studies will follow a randomized, double blinded, balanced, repeated measures design and the same protocol; except one will have an ad libitum pizza meal (study 1), while the other will have a fixed pizza meal (study 2) at 120 minutes. Half the participants will have blood drawn by IV and the other half will be finger prick.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoking males
* aged 20-30 years (min/max age)
* a body mass index between 20 and 25 kg/m2 (the range generally accepted as ideal/healthy by Health and Welfare Canada)

Exclusion Criteria:

* individuals diagnosed with diabetes
* those on medication
* breakfast skippers
* on an energy restricted diet
* this study excludes females because appetite and blood glucose during the female menstruation cycle changes due to fluctuations in hormones

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2017-10-21 (Actual); Study Completion 2017-10-21 (Actual)

PRIMARY OUTCOMES:
blood glucose | 0-200 minutes
  measured by finger prick blood samples by glucose meters

SECONDARY OUTCOMES:
appetite | 0-200 minutes
  measured by VAS questionnaire
satiety hormones | 0- 200mins
  measured by enzyme-linked immunosorbent assay (ELISA)
insulin | 0-200mins
  measured by ELISA
food intake | 120 minutes following consumption of the faba bean smoothie
  energy intake at ad-libitum pizza meal
physical comfort | 0-200 minutes
  measured by VAS questionnaire
energy/fatigue | 0-200 minutes
  measured by VAS questionaire

CONTACTS AND LOCATIONS:
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada